CLINICAL TRIAL: NCT03756974
Title: A Phase III, Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel-group Clinical Trial to Investigate the Efficacy and Safety of BX-1 for the Symptomatic Relief of Spasticity in Patients With Multiple Sclerosis (MS)
Brief Title: BX-1 in Spasticity Due to Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DroSpas-1
Record Dates: First submitted 2018-11-20; First posted 2018-11-28 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Spasticity Due to Multiple Sclerosis
Keywords: cannabinoid; dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BX-1 (dronabinol) (Experimental): BX-1
  Interventions: Drug: BX-1
- Placebo (Placebo Comparator): Placebo of BX-1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BX-1 — BX-1 (dronabinol), oral solution. All patients enrolled establish their individually tolerable dose by dose Titration.
  Arms: BX-1 (dronabinol)
Drug: Placebo — Placebo of BX-1, oral solution
  Arms: Placebo

SUMMARY:
To investigate the efficacy and safety of orally administered BX-1 compared to placebo in patients with spasticity due to multiple sclerosis not sufficiently controlled by current anti-spasticity medication

DETAILED DESCRIPTION:
The aim of the present phase III clinical trial is to demonstrate superiority of BX-1, an oral solution containing dronabinol, over placebo in patients with spasticity due to MS not sufficiently controlled by their current anti-spasticity medication.

The trial is designed to show that BX-1 is able to reduce spasticity in MS patients not showing sufficient response to their current anti-spasticity treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years
2. Presence of MS according to 2010 or 2017 revised McDonald criteria
3. Patients with stable MS for at least 3 months before enrolment in the opinion of the treating physician Note: Patients with a MS relapse during 3 month prior to enrolment are not considered to have stable MS
4. Ongoing spasticity for at least 3 months before enrolment
5. Spasticity in at least 2 lower limb muscles
6. Expanded Disability Status Scale (EDSS) score ≥ 3.0 and ≤ 6.5
7. Previous treatment with at least two different optimized oral MS anti-spasticity therapies before inclusion. Both treatment attempts must include at least baclofen or oral tizanidine, which can be combined with other anti-spasticity drugs.

   AND Patients currently receiving an optimized treatment corresponding to the last treatment attempt with stable dosage for at least 30 days prior to Visit 0.
8. Female patients of non-childbearing potential or if of childbearing potential using highly effective contraceptive methods or double barrier contraception.

   For men: no specific contraception methods need to be used.
9. Willingness to follow the study procedure for the whole duration of the trial and signed informed consent at screening prior to any trial-related procedure

Exclusion Criteria:

1. Any present disease other than MS that could affect spasticity (e.g. traumatic brain injury, spinal cord injury, brain damage due to a lack of oxygen, stroke, encephalitis, meningitis)
2. Intake of not permitted concomitant medication prior to screening and concomitant medication which should be unaltered prior to screening in an unstable dosage regimen
3. Significant fixed tendon contractures
4. History of epileptic seizures
5. History of or existing relevant CNS disorder (other than MS)
6. History of or existing relevant psychiatric disorders (e.g. schizophrenia, psychosis, manic disorders, severe depressive disorders, suicidal ideations, drug and/or alcohol abuse etc.)
7. Patients with a positive drug abuse screening test, except for medications used to treat a medical condition and reported as such by the patient; all patients with a positive result for cannabis/THC
8. History of or existing cardiac diseases or pathological findings (e.g. chronic insufficiency NYHA III/IV, severe arrhythmia, unstable angina pectoris, myocardial infarction within the past 6 months, QT prolongation)
9. Known HIV, and/or active Hepatitis B or C infection
10. History of or existing malignancy during the 5 years before screening except history of basal cell carcinoma and melanoma in situ
11. Significantly impaired renal function (estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1.73m2)
12. Significant impaired hepatic function (Alanine Aminotransferase > 3 times upper limit of normal or bilirubin > 2 times upper limit of normal, except Gilbert syndrome)
13. Known allergic reactions to the active ingredients used or to constituents of the IMP
14. Chronic or active infection requiring a systemic therapy
15. Pregnancy, breastfeeding or planned pregnancy
16. Any condition that interferes with the participation in the clinical trial at the discretion of the investigator
17. Patients not able to follow study instructions, not able to follow the study assessments defined by the protocol, unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial
18. Patients in custody by judicial or official order
19. Patients who are members of the staff of the trial centre, staff of the sponsor or CRO, the investigator him/herself or close relatives of the investigator
20. Parallel participation in another clinical trial, participation in another trial within less than 30 days or five half-lives of IMP (whatever is longer) to screening, or previous participation in this trial (except one time screening failures). A patient may be re-screened once, if any inclusion criterion is not met or any exclusion criterion is met during the first screening attempt.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Responder analysis: proportion of patients showing improvement in spasticity of 18% or more in average Numerical Rating Scale for Spasticity (NRS-S) assessment at end of treatment | 16 weeks
  Responder analysis: proportion of patients showing improvement in spasticity (change from baseline corresponding to the mean NRS-S score during 7 days prior to randomisation) of 18% or more in average NRS-S assessment at end of treatment (mean NRS-S score during 7 days prior to Visit 6).

SECONDARY OUTCOMES:
Responder analysis: proportion of patients showing improvement in spasticity (change from baseline) of 30% or more in average NRS-S assessment at end of treatment (Visit 6) | 16 weeks
Responder analysis: proportion of patients showing improvement in spasticity (change from baseline) of 50% or more in average NRS-S assessment at end of treatment (Visit 6) | 16 weeks
Time to response: time to reach first improvement in spasticity (change from baseline) of 18% or more, based on patient's daily spasticity assessment on the NRS-S | 16 weeks
Time to response: time to reach first improvement in spasticity (change from baseline) of 30% or more, based on patient's daily spasticity assessment on the NRS-S | 16 weeks
Weekly mean of the patient's daily spasticity assessments on the NRS-S during Visit 0 - Visit 6 | 21 weeks
Weekly mean of the patient's daily pain assessments on the Numerical Rating Scale for Pain (NRS-P) during Visit 0 - Visit 6 | 21 weeks
Responder analysis: proportion of patients showing improvement in pain (change from baseline) of 15% or more in average NRS-P assessment at end of treatment (Visit 6) | 16 weeks
Responder analysis: proportion of patients showing improvement in pain (change from baseline) of 30% or more in average NRS-P assessment at end of treatment (Visit 6) | 16 weeks
Time to response: time to reach first improvement in pain (change from baseline) of 15% or more, based on patient's pain assessment on the NRS-P | 16 weeks
Time to response: time to reach first improvement in pain (change from baseline) of 30% or more, based on patient's pain assessment on the NRS-P | 16 weeks
Weekly mean of the patient's daily spasm frequency and severity assessments on the Penn Spasm Frequency Scale (PSFS) during Visit 0 - Visit 6 | 21 weeks
Mean change from baseline of spasm frequency and severity assessments on the PSFS at end of treatment (Visit 6) | 16 weeks
Mean change from baseline of Timed 25-Foot Walk (T25-FW) at Visit 4 and Visit 6 | 16 weeks
Responder analysis: proportion of patients showing improvement in TF25-FW (change from baseline) of 20% or more at Visit 6 | 16 weeks
Mean change from baseline of the physical and psychological impact of multiple sclerosis assessed with the Multiple Sclerosis Impact Scale- 29 version 2 (MSIS-29 v2) at Visit 4 and Visit 6 | 16 weeks
Mean change from baseline of quality of life measured with Short-Form Health Survey of the Medical Outcomes Study Version 2 (SF-36 v2) at Visit 6 | 16 weeks
Mean change from baseline of sleep quality measured with the Numerical Rating Scale for Sleep Quality (NRS-SQ) at Visit 3 - Visit 6 | 12 weeks
Mean change from baseline of fatigue measured with the Numerical Rating Scale for Fatigue (NRS-F) at Visit 3 - Visit 6 | 12 weeks
Overall patients' status measured by Patient´s Global Impression of Change scale (PGIC) at Visit 5 and Visit 6 | 16 weeks
Overall patients' status measured by Clinical Global Impression - Improvement scale (CGI-I) at Visit 5 and Visit 6 | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luitgard Spitznagel-Schminke, Study Director — Bionorica SE
Locations (30):
- Czechia (8):
  - Investigative Site, Choceň
  - Investigative Site, Havířov
  - Investigative Site, Hradec Králové
  - Investigative site, Hradec Králové
  - Investigative Site, Olomouc
  - Investigative Site, Pilsen
  - Investigative Site, Prague
  - Investigative Site, Teplice
- Germany (2):
  - Investigative Site, Freiburg im Breisgau
  - Investigative Site, Ulm
- Hungary (7):
  - Investigative Site, Budapest
  - Investigative Site, Debrecen
  - Investigative Site, Győr
  - Investigative Site, Miskolc
  - Investigative Site, Szeged
  - Investigative Site, Szolnok
  - Investigative Site, Tatabánya
- Poland (7):
  - Investigative Site, Bydgoszcz
  - Investigative Site, Częstochowa
  - Investigative Site, Katowice
  - Investigative Site, Krakow
  - Investigative Site, Plewiska
  - Investigative Site, Poznan
  - Investigative Site, Warsaw
- Spain (6):
  - Investigative Site, Barcelona
  - Investigative Site, L'Hospitalet de Llobregat
  - Investigative Site, Madrid
  - Investigative Site, Málaga
  - Investigative Site, Salt
  - Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: No